CLINICAL TRIAL: NCT05315128
Title: Intralesional Methotrexate Versus Intramuscular Methotrexate in the Treatment of Non-melanoma Skin Cancers
Brief Title: Intralesional Versus Intramuscular Methotrexate for Non-melanoma Skin Cancers
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Zagazig University (Other Government)
Responsible Party: Principal Investigator, Basma Magdy Elkholy, MD, Dr, Zagazig University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: IRB# 6029/-6-7-2020
Record Dates: First submitted 2022-02-15; First posted 2022-04-07 (Actual); Last update posted 2022-04-07 (Actual); Status verified 2022-04

CONDITIONS: Non-melanoma Skin Cancers
Keywords: Non-melanoma skin cancer; Intralesional methotrexate; Systemic methotrexate; Intramuscular methotrexate; Keratoacanthoma; Basal cell carcinoma; Squamous cell carcinoma
MeSH Terms: conditions — Keratoacanthoma; Carcinoma, Basal Cell; Carcinoma, Squamous Cell | interventions — Methotrexate

STUDY DESIGN:
Who Masked: Participant, Care Provider
Masking Description: Double-blinded
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intralesional methotrexate (Active Comparator): Group A 30 patients received intralesional injection of MTX with an insulin syringe into the tumor at a dose ranging between 12.5 mg to 25 mg according to the tumor size every week until complete improvement or for a maximum of 8 sessions.
  Interventions: Drug: Methotrexate
- Intramuscular methotrexate (Active Comparator): Group B 30 patients received systemic MTX (SC, or IM) was injected at a dose of 25 mg every week until clearance or for a maximum of 8 sessions.
  Interventions: Drug: Methotrexate

INTERVENTIONS:
Drug: Methotrexate — A randomized comparative effectiveness clinical trial

SUMMARY:
to compare the effectiveness and safety of intralesional vs. systemic MTX in NMSC management

DETAILED DESCRIPTION:
Intralesional methotrexate (MTX) could to be promising conservative alternative for non-melanoma skin cancer (NMSC). Systemic MTX was attempted as adjuvant for locally-advanced NMSC.

ELIGIBILITY:
Inclusion Criteria:

• Adult patients of both sexes with histologically-confirmed primary or recurrent non- metastatic NMSCs of different types (BCC,SCC, and/or KA), sites, number, sizes and duration were included in the study.

Exclusion Criteria:

• Hypersensitivity reactions to methotrexate, liver or kidney disease, immunosuppressive conditions, HIV, HBV, and HCV infection, hematological abnormalities and metastasis. Pregnant or lactating women, females in their child-bearing period not using or refusing contraceptive methods, and those who had any other form of NMSC management in the month preceding enrollment.

Ages: 20 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2020-07-06 (Actual); Primary Completion 2021-08-10 (Actual); Study Completion 2021-12-06 (Actual)

PRIMARY OUTCOMES:
Reduction in size and number of tumors | up to 1 month after the last session
  Patients were divided into 3 groups: responders (if the tumor has regressed by > 50%), partial responders (tumor regression < 50%), and non- responders (no improvement at all or worsening).

SECONDARY OUTCOMES:
Adverse effects | Starting from the first session and up to 6-months after the last session
Recurrence | till the end of follow up duration (6 months)
  after achieving response greater than 50% of the tumor
New NMSC lesions elsewhere | from the start of the study and till the end of follow up period (6 months)

CONTACTS AND LOCATIONS:
Locations (1):
- Zagazig university, Zagazig, Sharqia Province, Egypt

IPD SHARING:
Plan to Share IPD: Undecided